





# Development and Evaluation of a Psychomotor Rehabilitation Nursing Plan for the Elderly with Mild Cognitive Impairment to Promote Cognitive Health

February 2025

Protocol ID: JZMULL2025230

Ethics Approval Number: USM/JEPeM/PP/24090806

<u>CONTOH</u> <u>ATTACHMENT B</u>

## RESEARCH INFORMATION

Research Title: Development and Evaluation of a Psychomotor Rehabilitation Nursing Plan for the Older

Adults with Cognitive Impairment to Promote Cognitive Health

#### Name of main and co-Researcher:

Main researcher: Wang Ying (China Health Professional Qualification no. for nursing: 2017121702320300001; China Health Professional Qualification no. for rehabilitation: 3022022072107022)

Co-researcher / Supervisor : Dr. Noor Mastura Binti Mohd Mujar (GCP no. 841129-08-5022)

#### INTRODUCTION

With the aging of the population, the number of older adults with mild cognitive impairment (MCI) has increased year by year, which has caused serious social and family burdens. At present, the existing drug treatment effect is limited. Studies show the application value of non-drug treatment in the older adults with mild cognitive impairment.

You (your family) are invited to take part voluntarily in an interventional research. This research is about to investigate a psychomotor rehabilitation nursing intervention plan to promote cognitive performance in older adults.

It is important that you read and understand this research information before agreeing to participate in this study. You will receive a copy of this form to keep for your records if you agree to participate.

Your participation in this study is expected to 3 months. This study is estimated to include up to 76 participants.

# **PURPOSE OF THE STUDY**

The purpose of this study is to determine whether a PMT rehabilitation nursing plan is effective in improving the cognitive status of older adults.

#### **PARTICIPANTS CRITERIA**

The research team members will discussed your eligibility to participate in this study. It is important that you are completely truthful with the staff including your health history.

Inclusion criteria: 1. Older adults are aged 50 years and above. 2. Subjective cognitive complaints from the individual or caregiver. 3. Screening for MCI using the Mini-Cog scores between 0-2. 4. Basic language communication, listening, speaking, and understanding skills. 5. Ability to provide informed consent.

Exclusion criteria: 1. Diagnosed with severe psychiatric conditions (e.g., schizophrenia, major depressive disorder). 2. It is at the end stage of important functional organ diseases, such as malignant tumors, cardiac failure, etc. 3. Limb dysfunction. 4. Diagnosed with dementia.

Withdrawal criteria: 1. Withdrawal of consent by the participant. 2. Non-compliance with study requirements (e.g., missing >25% sessions). 3. Significant health deterioration affecting participation.

### **STUDY PROCEDURES**

Older adults will be engaged in a 12-week PMT rehabilitation nursing plan involving 2 phases of relaxation and breathing exercises, face exercises, hand exercises and mind exercises to promote cognitive health. Phase 1 (Weeks 1-6): Includes relaxation and breathing exercises (10 minutes), facial exercises (10 minutes), bead maze activities (10 minutes), geometric shape puzzles (10 minutes), and finger exercises (20 minutes). Phase 2 (Weeks 7-12): Includes relaxation and breathing exercises (10 minutes), Tai Chi ball exercises (10 minutes), screw and nut assembly activities (10 minutes), tangram puzzles (10 minutes), and

upper limb music exercises (20 minutes). The experimental group will be given interventions, twice a week every Tuesday and Thursday 9-10 am along with the study intervention. Meanwhile, the control group will be given a standard health education on cognitive health.

I will use a questionnaire to assess cognitive status. First, I will collect some personal and social information from you. There are 7 questions in total, which will take no more than 5 minutes. Then, I will conduct questionnaire surveys before the intervention (baseline) and after the intervention (12 weeks). The questionnaires involved include MoCA, which has 11 questions and takes about 10 minutes; PANSS, which has 30 questions and takes about 20 minutes; HAMA-14, which has 14 questions and takes about 10 minutes; HAMD-17, which has 17 questions and takes about 15 minutes. All questionnaires will take no more than 60 minutes.

Participants are required to attend the intervention sessions on time, undergo regular cognitive assessments, and provide necessary health information and feedback. Participants are expected to cooperate with the research team and follow the study protocol.

#### RISKS

- 1. Fall or Injury Risk: Older adults may have weaker muscle strength, balance, and coordination, which makes them more prone to falls or injuries during rehabilitation activities. If participants fall or are injured during the intervention, necessary medical support will be provided.
- 2. Feelings of Frustration: If older adults do not experience the expected progress during rehabilitation, they may develop feelings of frustration, disappointment, or reduced self-efficacy. If participants experience any discomfort, psychological support will be provided, and they may withdraw from the study at any time.

#### REPORTING HEALTH EXPERIENCES.

Please contact, at any time, the following researcher if you experience any health problem either directly or indirectly related to this study.

Wang Ying [China Health Professional Qualification no. for nursing: 2017121702320300001; China Health Professional Qualification no. for rehabilitation: 3022022072107022] at hone No. +86 18640669145>.

#### PARTICIPATION IN THE STUDY

- 1. Your taking part in this study is entirely voluntary. You may refuse to take part in the study or you may stop your participation in the study at anytime, without any penalty or loss of benefits to which you are otherwise entitled.
- 2. Your participation also may be stopped by the research team without your consent if in any form you have violated the study eligibility criteria. The research team member will discussed with you if the matter arises
- 3. Participants will be compensated for any medical expenses related to study interventional-related injuries, and all healthcare costs incurred due to study interventional-related events will be covered by the research team
- 4. If the participant experiences disability or death due to a study interventional-related injury, the participant or their family will receive appropriate compensation as per the study's legal coverage.

#### POSSIBLE BENEFITS [Benefit to Individual, Community, University]

- 1. This study finding may benefit older adults who live in care institutions, rehabilitation hospitals, communities, and families to improve physical function and promote cognitive function.
- 2. It can lower societal healthcare costs and long-term caregiving expenses and help delay the health decline of older adults, assisting society in addressing the health and economic challenges an aging population poses.
- 3. Older adults' participation in this study provides universities with important research subjects, advancing academic research, particularly in geriatric medicine, rehabilitation medicine, psychology, and nursing, and promoting the development and application of innovative intervention programs.
- 4. You will not recieve any compensation from this study. However you may get reimbursement for your travelling cost while in the study duration.
- 5. If the study intervention is proven safe and effective, participants will be given the opportunity to continue receiving the intervention after the study concludes.

#### **QUESTIONS**

If you have any question about this study or your rights, please contact;

If you have any questions regarding the Ethical Approval or any issue / problem related to this study, please contact:

Mr. Mohd Bazlan Hafidz Mukrim Secretary of Human Research Ethics Committee USM Division of Research & Innovation (R&I) USM Health Campus

Tel. No.: 09-767 2354 / 09-767 2362

Email: bazlan@usm.my

OR

Miss Nor Amira Khurshid Ahmed Secretariat of Human Research Ethics Committee USM Research Creativity & Management Office (RCMO) USM Main Campus, Penang

Tel. No.: 04-6536537

Email: noramira@usm.my

#### CONFIDENTIALITY

- **1.** Your information and study data will be kept confidential by the researchers and will not be made publicly available unless disclosure is required by law. At the end of the study, all personally identifiable information will be destroyed, and remaining data will be stored anonymously for future analysis.
- 2. Data obtained from this study that does not identify you individually will be published for knowledge purposes. Upon completion of the study, all participants will receive a summary report of the study findings, including any health-related recommendations.
- 3. Your original records may be reviewed by the researcher, the Ethical Review Board for this study, and regulatory authorities for the purpose of verifying the study procedures and/or data. Your information may be held and processed on a computer. Only research team members are authorized to access your information. Participants have the right to access their study-related records at any time, including health assessments and intervention progress reports.

# **OTHER**

The investigator in this study serves as an investigator and the services provider for the study intervention.

By signing this consent form, you authorize the record review, information storage and data process described above.

#### **SIGNATURES**

To be entered into the study, you or a legal representative must sign and data the signature page [ATTACHMENT S and ATTACHMENT P]

# Subject Information and Consent Form (Signature Page)

Research Title: Development and Evaluation of a Psychomotor Rehabilitation Nursing Plan

for the Older Adults with Cognitive Impairment to Promote Cognitive Health

**Researcher's Name :** Wang Ying (China Health Professional Qualification no. for nursing: 2017121702320300001; China Health Professional Qualification no. for rehabilitation: 3022022072107022)

Co-researcher / Supervisor: Dr. Noor Mastura Binti Mohd Mujar(GCP no. 841129-08-5022

To become a part this study, you or your legal representative must sign this page. By signing this page, I am confirming the following:

- I have read all of the information in this Patient Information and Consent Form including any information regarding the risk in this study and I have had time to think about it.
- All of my questions have been answered to my satisfaction.
- I voluntarily agree to be part of this research study, to follow the study procedures, and to provide necessary information to the doctor, nurses, or other staff members, as requested.
- I may freely choose to stop being a part of this study at anytime.
- I have received a copy of this Participant Information and Consent Form to keep for myself.

| Participant Name | |
|-------------------------------------------------------|-----------------|
| Participant I.C No | |
| Signature of Participant or Legal Representative | Date (dd/MM/yy) |
| Name of Individual Conducting Consent Discussion | |
| Signature of Individual Conducting Consent Discussion | Date (dd/MM/yy) |
| Name & Signature of Witness | Date (dd/MM/yy) |

Note: i) All participants who are involved in this study will not be covered by insurance.

# Participant's Material Publication Consent Form Signature Page

Research Title: Development and Evaluation of a Psychomotor Rehabilitation Nursing Plan

for the Older Adults with Cognitive Impairment to Promote Cognitive Health

Researcher's Name: Wang Ying (China Health Professional Qualification no. for nursing: 2017121702320300001; China Health Professional Qualification no. for rehabilitation:

3022022072107022)

Co-researcher / Supervisor: Dr. Noor Mastura Binti Mohd Mujar(GCP no. 841129-08-5022)

To become a part this study, you or your legal representative must sign this page.

By signing this page, I am confirming the following:

- I understood that my name will not appear on the materials published and there have been efforts to make sure that the privacy of my name is kept confidential although the confidentiality is not completely guaranteed due to unexpected circumstances.
- I have read the materials or general description of what the material contains and reviewed all photographs and figures in which I am included that could be published.
- I have been offered the opportunity to read the manuscript and to see all materials in which I am included, but have waived my right to do so.
- All the published materials will be shared among the medical practitioners, scientists and journalist world wide.
- The materials will also be used in local publications, book publications and accessed by many local and international doctors world wide.
- I hereby agree and allow the materials to be used in other publications required by other publishers with these conditions:
- The materials will not be used as advertisement purposes nor as packaging materials.
- The materials will not be used out of contex i.e.: Sample pictures will not be used in an article which is unrelated subject to the picture.

| Participant Name | | |
|-------------------------|-------------------------|-----------------|
| <br>Participant I.C No. | Participant's Signature | Date (dd/MM/yy) |
| Name and Signature of I | | Date (dd/MM/yy) |

Note: i) All participants who are involved in this study will not be covered by insurance.

# **APPENDICES**

# **Data Collection Form**

| Name: | ID: |
|---|---|
| Elderly's General information | 1: |
| 1.Sex | |
| -Female | : |
| -Male | : |
| 2.Age (years) | : |
| 3.Education Level | |
| -Illiteracy | : |
| -Primary school | : |
| -Middle school | : |
| -College or above | : |
| 4. Family history of dementia ( | Yes or No ) : |
| 5. Marital status | |
| -Single / Divorced / Wido | owed : |
| -Married | : |
| 6.Personal annual income | : |
| 7. Chronic disease (Yes or No. 1 | f yes, please write the specific disease name) |

MONTREAL COGNITIVE ASSESSMENT (MOCA) Version 7.1 Original Version

NAME: Education: Sex:

Date of birth : DATE :

| VISUOSPATIAL / E E End S Begin | (A) (B) (2) (4) (3) | | | Copy<br>cube | Draw<br>(3 poin | | Ten past elev | en) | POINTS |
|---|---|---|---|---|---|---|---|---|---|
| © | [ ] | | | [ ] | [ ]<br>Contou | [<br>r Nu | - | [ ]<br>Hands | /5 |
| NAMING | | | | | E STAN | | | | /3 |
| MEMORY repeat them. Do 2 trial Do a recall after 5 minu | Read list of words, subject<br>s, even if 1st trial is successful.<br>utes. | must 1st tri 2nd tri | | VELVE | т сн | URCH | DAISY | RED | No<br>points |
| ATTENTION | Read list of digits (1 digit/ | | has to repeat t | | | | [ ] 2 1 8 | | /2 |
| Read list of letters. The | subject must tap with his h | and at each letter | | | LBAFAI | KDEAA | AJAMOF | A A B | /1 |
| Serial 7 subtraction sta | arting at 100 | | ] 86<br>rect subtractions: | [ ] 79<br><b>3 pts</b> , 2 or | | [ ] 72<br><b>pts</b> , 1 corr | [ ]<br>ect: <b>1 pt</b> , 0 corre | | /3 |
| LANGUAGE | Repeat : I only know that<br>The cat always I | | help today. [ | ] | | | • | | /2 |
| Fluency / Name | maximum number of words | in one minute that | begin with the | letter F | | []_ | (N ≥ 11 w | ords) | /1 |
| ABSTRACTION | Similarity between e.g. bar | nana - orange = fru | it []tr | ain – bicycl | le [ ] | watch - rı | uler | | /2 |
| DELAYED RECALL | Has to recall words WITH NO CUE | | | | DAISY<br>[ ] | RED<br>[ ] | Points for<br>UNCUED<br>recall only | | /5 |
| Optional | Category cue<br>Multiple choice cue | | | | | | | | |
| ORIENTATION | [ ] Date [ ] | Month [ | ] Year | [ ] Day | [ | ] Place | [ ] Ci | ty | /6 |
| © <b>Z.Nasreddine MI</b> Administered by: | , | www.mocate | est.org | Normal | ≥26 / 30 | 1017 | L<br>Add 1 point if | _<br>≤ 12 yr edu | _/30 |

| POSITIVE AND NEGATIVE SYNDROME SCALE (PANSS) | |
|---|---|
| ITEMS | SCORE |
| POSITIVE SCALE (P): | |
| P1. DELUSIONS - Beliefs which are unfounded, unrealistic and idiosyncratic. | |
| P2. CONCEPTUAL DISORGANISATION - Disorganized process of thinking characterized by disruption of goal-directed sequencing, e.g. circumstantiality, loose associations, tangentiality, gross illogicality or thought block. | |
| P3. HALLUCINATORY BEHAVIOUR - Verbal report or behavior indicating perceptions that are not generated by external stimuli. These may occur in the auditory, visual, olfactory, or somatic realms. | |
| P4. EXCITEMENT - Hyperactivity as reflected in accelerated motor behavior, heightened responsivity to stimuli, hypervigilance or excessive mood lability. | |
| P5. GRANDIOSITY - Exaggerated self-opinion and unrealistic convictions of superiority, including delusions of extraordinary abilities, wealth, knowledge, fame, power and moral righteousness. | |
| P6. SUSPICIOUSNESS/PERSECUTION - Unrealistic or exaggerated ideas of persecution, as reflected in guardedness, ad distrustful attitude, suspicious hypervigilance or frank delusions that others mean harm. | |
| P7. HOSTILITY - Verbal and nonverbal expressions of anger and resentment, including sarcasm, passive-aggressive behavior, verbal abuse, and assualtiveness. | |
| NEGATIVE SCALE (N): | |
| N1. BLUNTED AFFECT - Diminished emotional responsiveness as characterized by a reduction in facial expression, modulation of feelings and communicative gestures. | |
| N2. EMOTIONAL WITHDRAWAL - Lack of interest in, involvement with, and affective commitment to life's events. | |
| N3. POOR RAPPORT - Lack of interpersonal empathy, openness in conversation and sense of closeness, interest or involvement with the interviewer. This is evidenced by interpersonal distancing and reduced verbal and nonverbal communication | |
| N4. PASSIVE/APATHETIC SOCIAL WITHDRAWAL - Diminished interest and initiative in social interactions due to passivity, apathy, anergy or avolition. This leads to reduced interpersonal involvements and neglect of activities of daily living. | |
| N5. DIFFICULTY IN ABSTRACT THINKING - Impairment in the use of the abstract-symbolic mode of thinking, as evidenced by difficulty in classification, forming generalizations, and proceeding beyond concrete or egocentric thinking in problem-solving tasks. | |
| N6. LACK OF SPONTANEITY AND FLOW OF CONVERSATION - Reduction in the normal flow of communication associated with apathy, avolition, defensiveness or cognitive deficit. This is manifested by diminished fluidity and productivity of the verbal interactional process. | |
| N7. STEREOTYPED THINKING - Decreased fluidity, spontaneity and flexibility of thinking, as evidenced in rigid, repetitious or barren thought content. | |

| GENERAL PSYCHOPATHOLOGY SCALE(G): | |
|---|---|
| G1. SOMATIC CONCERN - Physical complaints or beliefs about bodily illness or malfunctions. This may range from a vague sense of ill being to clear-cut delusions of catastrophic physical disease. | |
| G2. ANXIETY - Subjective experience of nervousness, worry, apprehension or restlessness, ranging from excessive concern about the present or future to feelings of panic. | |
| G3. GUILT FEELINGS - Sense of remorse or self-blame for real or imagined misdeeds in the past. | |
| G4. TENSION -Overt physical manifestations of fear, anxiety, and agitation, such as stiffness, tremor, profuse sweating and restlessness. | |
| G5. MANNERISMS AND POSTURING – Unnatural movements or posture as characterized be an awkward, stilted, disorganised, or bizarre appearance. | |
| G6. DEPRESSION - Feelings of sadness, discouragement, helplessness and pessimism. | |
| G7. MOTOR RETARDATION – Reduction in motor activity as reflected in slowing or lessening or movements and speech, diminished responsiveness of stimuli, and reduced body tone. | |
| G8. UNCOOPERATIVENESS - Active refusal to comply with the will of significant others, including the interviewer, hospital staff or family, which may be associated with distrust, defensiveness, stubbornness, negativism, rejection of authority, hostility or belligerence. | _ |
| G9. UNUSUAL THOUGHT CONTENT - Thinking characterized by strange, fantastic, or bizarre ideas, ranging from those that are remote or atypical to those that are distorted, illogical, and patently absurd. | |
| G10. DISORIENTATION - Lack of awareness of one's relationship to the milieu, including persons, place and time, which may be due to confusion or withdrawal. | |
| G11. POOR ATTENTION - Failure in focused alertness manifested<br>by poor concentration, distractibility from internal and external<br>stimuli, and difficulty in harnessing, sustaining or shifting focus to<br>new stimuli. | |
| G12. LACK OF JUDGEMENT AND INSIGHT - Impaired awareness or understanding of one's own psychiatric condition and life situation. This is evidenced by failure to recognize past or present psychiatric illness or symptoms, denial of the need for psychiatric hospitalization or treatment, decisions characterized by poor anticipation or consequences, and unrealistic short-term and long-range planning. | |
| G13. DISTURBANCE OF VOLITION – Disturbance in the wilful initiation, sustenance, and control of one's thoughts, behavior, movements, and speech. | |
| G14. POOR IMPULSE CONTROL - Disordered regulation and control of action on inner urges, resulting in sudden, unmodulated, arbitrary or misdirected discharge of tension and emotions without concern about consequences. | |
| G15. PREOCCUPATION - Absorption with internally generated thoughts and feelings and with autistic experiences to the detriment of reality orientation and adaptive behavior. | |
| G16. ACTIVE SOCIAL AVOIDANCE - Diminished social involvement associated with unwarranted fear, hostility, or distrust. | |

# **HAMILTON ANXIETY RATING SCALE (HAM-A)**

Below is a list of phrases that describe certain feelings that people have. Rate the patients by finding the answer that best describes the extent to which he/she has these conditions. Select one of the five responses for each of the 14 questions.

| | 0 =<br>Not<br>present | 1 =<br>Mild | 2 =<br>Moderate | 3 =<br>Severe | 4 =<br>Very<br>severe |
|---|---|---|---|---|---|
| 1. Anxious mood Worries, anticipation of the worst, fearful anticipation, irritability. | | | | | |
| 2. Tension Feelings of tension, fatigability, startle response, moved to tears easily, trembling, feelings of restlessness, inability to relax. | | | | | |
| 3. Fears Of dark, of strangers, of being left alone, of animals, of traffic, of crowds. | | | | | |
| 4. Insomnia Difficulty in falling asleep, broken sleep, unsatisfying sleep<br>and fatigue on waking, dreams, nightmares, night terrors. | | | | | |
| 5. Intellectual Difficulty in concentration, poor memory. | | | | | |
| <b>6. Depressed mood</b> Loss of interest, lack of pleasure in hobbies, depression, early waking, diurnal swing. | | | | | |
| 7. Somatic (muscular) Pains and aches, twitching, stiffness, myoclonic jerks, grinding of teeth, unsteady voice, increased muscular tone. | | | | | |
| <ol> <li>Somatic (sensory) Tinnitus, blurring of vision, hot and cold flushes, feelings of<br/>weakness, pricking sensation.</li> </ol> | | | | | |
| <ol> <li>Cardiovascular symptoms Tachycardia, palpitations, pain in chest, throbbing of vessels, fainting feelings, missing beat.</li> </ol> | | | | | |
| Respiratory symptoms Pressure or constriction in chest, choking feelings, sighing, dyspnea. | | | | | |
| 11. Gastrointestinal symptoms Difficulty in swallowing, wind abdominal pain, burning sensations, abdominal fullness, nausea, vomiting, borborygmi, looseness of bowels, loss of weight, constipation. | | | | | |
| 12. Genitourinary symptoms Frequency of micturition, urgency of micturition, amenorrhea, menorrhagia, development of frigidity, premature ejaculation, loss of libido, impotence. | | | | | |
| 13. Autonomic symptoms Dry mouth, flushing, pallor, tendency to sweat, giddiness, tension headache, raising of hair. | | | | | |
| 14. Behaviour at interview Fidgeting, restlessness or pacing, tremor of hands, furrowed brow, strained face, sighing or rapid respiration, facial pallor, swallowing, etc. | | | | | |

Scoring: Each item is scored on a scale of 0 (not present) to 4 (very severe), with a total score range of 0–56, where <17 indicates mild severity, 18–24 mild to moderate severity, 25–30 moderate to severe and 31-56 severe to very severe.

Copyright notice: The HAM-A is in the public domain.

References: 1. Hamilton M.The assessment of anxiety states by rating. Br J Med Psychol 1959;32:50-5. 2. Maier W, Buller R, Philipp M, Heuser I. The Hamilton Anxiety Scale: reliability, validity and sensitivity to change in anxiety and depressive disorders. J Affect Disord 1988;14(1):61-8. 3. Borkovec T and Costello E. Efficacy of applied relaxation and cognitive behavioral therapy in the treatment of generalized anxiety disorder. J Clin Consult Psychol 1993;61(4):611-9.

#### HAMILTON DEPRESSION RATING SCALE (HAM-D17)

| | TIAMILI ON BEI RESSION | MATING SCALE (HAMI-DIT) |
|---|---|---|
| 1 | DEPRESSED MOOD (sadness, hopeless, helpless, worthless) | 10 ANXIETY PSYCHIC |
| | 0 _ Absent. | 0 No difficulty. |
| | I _ These feeling states indicated only on questioning. | I Subjective tension and irritability. |
| | 2 These feeling states spontaneously reported verbally. | <ol> <li>Worrying about minor matters.</li> </ol> |
| | 3 Communicates feeling states non-verbally, i.e. through | 3 Apprehensive attitude apparent in face or speech. |
| | facial expression, posture, voice and tendency to weep. | 4 Fears expressed without questioning. |
| | 4 _ Patient reports virtually only these feeling states in | |
| | his/her spontaneous verbal and non-verbal | II ANXIETY SOMATIC (physiological concomitants of |
| | communication. | anxiety) such as: |
| 2 | FEELINGS OF GUILT | gastro-intestinal – dry mouth, wind, indigestion, diarrhea, |
| 2 | 0 Absent. | cramps, belching |
| | Self reproach, feels he/she has let people down. | cardio-vascular - palpitations, headaches |
| | 2 Ideas of guilt or rumination over past errors or sinful | respiratory – hyperventilation, sighing |
| | deeds. | urinary frequency |
| | 3 Present illness is a punishment. Delusions of guilt. | sweating |
| | 4 Hears accusatory or denunciatory voices and/or | 0 Absent. |
| | experiences threatening visual hallucinations. | I _ Mild. |
| | experiences un eatening visual nandemations. | 2 Moderate. |
| 3 | SUICIDE | 3 Severe. |
| | 0 Absent. | 4 Incapacitating. |
| | I Feels life is not worth living. | IS COMMITTED COMPTONE CASTRO INTESTIMAL |
| | 2 _ Wishes he/she were dead or any thoughts of possible | 12 SOMATIC SYMPTOMS GASTRO-INTESTINAL |
| | death to self. | 0 _ None. |
| | 3 Ideas or gestures of suicide. | _ Loss of appetite but eating without staff |
| | 4 _ Attempts at suicide (any serious attempt rate 4). | encouragement. Heavy feelings in abdomen. |
| | | 2 _ Difficulty eating without staff urging. Requests or |
| 4 | INSOMNIA: EARLY IN THE NIGHT | requires laxatives or medication for bowels or |
| | 0 No difficulty falling asleep. | medication for gastro-intestinal symptoms. |
| | Complains of occasional difficulty falling asleep, i.e. | 13 GENERAL SOMATIC SYMPTOMS |
| | more than ½ hour. | |
| | 2 Complains of nightly difficulty falling asleep. | 0 _ None. I Heaviness in limbs, back or head. Backaches, |
| | | ·—· |
| 5 | INSOMNIA: MIDDLE OF THE NIGHT | headaches, muscle aches. Loss of energy and |
| | 0 No difficulty. | fatigability. |
| | I _ Patient complains of being restless and disturbed | 2 _ Any clear-cut symptom rates 2. |
| | during the night. | 14 GENITAL SYMPTOMS (symptoms such as loss of libido, |
| | 2 Waking during the night – any getting out of bed rates | menstrual disturbances) |
| | 2 (except for purposes of voiding). | 0 Absent. |
| | | I Mild. |
| 6 | INSOMNIA: EARLY HOURS OF THE MORNING | 2 Severe. |
| | 0 _ No difficulty. | Z _ Severe. |
| | Waking in early hours of the morning but goes back | 15 HYPOCHONDRIASIS |
| | to sleep. | 0 Not present. |
| | 2 Unable to fall asleep again if he/she gets out of bed. | I Self-absorption (bodily). |
| 7 | WORK AND ACTIVITIES | 2 Preoccupation with health. |
| , | | 3 Frequent complaints, requests for help, etc. |
| | No difficulty. I Thoughts and feelings of incapacity, fatigue or | 4 Hypochondriacal delusions. |
| | I Thoughts and feelings of incapacity, fatigue or weakness related to activities, work or hobbies. | |
| | 2 Loss of interest in activity, hobbies or work – either | 16 LOSS OF WEIGHT (RATE EITHER a OR b) |
| | directly reported by the patient or indirect in | a) According to the b) According to weekly |
| | listlessness, indecision and vacillation (feels he/she has | patient: measurements: |
| | to push self to work or activities). | 0 No weight loss. 0 Less than I lb weight loss in |
| | Decrease in actual time spent in activities or decrease | week. |
| | in productivity. Rate 3 if the patient does not spend at | I _ Probable weight I _ Greater than I lb weight loss |
| | least three hours a day in activities (job or hobbies) | loss associated with in week. |
| | excluding routine chores. | present illness. |
| | 4 _ Stopped working because of present illness. Rate 4 if | 2 Definite (according 2 Greater than 2 lb weight loss |
| | patient engages in no activities except routine chores, | to patient) weight in week. |
| | or if patient fails to perform routine chores unassisted. | loss. |
| 8 | RETARDATION (slowness of thought and speech, impaired | |
| | lity to concentrate, decreased motor activity) | 17 INSIGHT |
| | 0 Normal speech and thought. | 0 Acknowledges being depressed and ill. |
| | I Slight retardation during the interview. | I Acknowledges illness but attributes cause to bad food, |
| | 2 Obvious retardation during the interview. | climate, overwork, virus, need for rest, etc. |
| | 3 Interview difficult. | 2 Denies being ill at all. |
| | 4 Complete stupor. | |
| | | Total score: _ |
| 9 | AGITATION | |
| | 0 None. | |
| | I Fidgetiness. | |
| | 2 Playing with hands, hair, etc. | |
| | 3 Moving about, can't sit still. | |
| | 4 Hand wringing, nail biting, hair-pulling, biting of lips. | |

Ratings should be based upon symptoms over the past <u>one week</u>.

Ratings should be based on a clinical interview, supplemented, where necessary, by collateral history from caregivers. Hamilton, M. (1960). A rating scale for depression. *Journal of Neurology, Neurosurgery, and Psychiatry*, 23(1), 56–62. https://doi.org/10.1136/jnnp.23.1.56